CLINICAL TRIAL: NCT03231917
Title: Water Immersion and Polyp Detection: A Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: White River Junction Veterans Affairs Medical Center (U.S. Federal Agency)
Collaborators: Indiana University (Other)
Responsible Party: Principal Investigator, Joseph Anderson, Associate Professor, White River Junction Veterans Affairs Medical Center
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Screening
Other Study IDs: 1000344-1
Record Dates: First submitted 2017-07-25; First posted 2017-07-27 (Actual); Results first posted 2019-07-12 (Actual); Last update posted 2019-07-12 (Actual); Status verified 2019-04

CONDITIONS: Adenoma; Colonic Neoplasms
MeSH Terms: conditions — Adenoma; Colonic Neoplasms

STUDY DESIGN:
Intervention Model Description: In one randomized group, water infusion will be employed as the first method for mucosal inspection while in a second group, CO2 insufflation will be used first. This study will be different than usual care since the participants will receive two successive or tandem colonoscopies versus one
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Water Infusion first (Experimental): In this group patients will receive a colonoscopy with water infusion for mucosal inspection and then receive a colonoscopy with CO2 insufflation.
  Interventions: Procedure: Water Infusion first
- CO2 Insufflation First (Experimental): In this group patients will receive a colonoscopy with CO2 insufflation for mucosal inspection and then receive a colonoscopy with water infusion.
  Interventions: Procedure: CO2 Insufflation First

INTERVENTIONS:
Procedure: Water Infusion first — In this group patients will receive a colonoscopy with water infusion for mucosal inspection and then receive a colonoscopy with CO2 insufflation.
  Arms: Water Infusion first
Procedure: CO2 Insufflation First — In this group patients will receive a colonoscopy with CO2 insufflation for mucosal inspection and then receive a colonoscopy with water infusion .
  Arms: CO2 Insufflation First

SUMMARY:
We plan to conduct a randomized trial of tandem colonoscopies comparing water infusion and air insufflation for inspection of mucosa on withdrawal. In one randomized group, water infusion will be employed as the first method for mucosal inspection while in a second group, CO2 insufflation will be used first. This study will be different than usual care since the participants will receive two successive or tandem colonoscopies versus one

ELIGIBILITY:
Inclusion Criteria:

* all adults 50 years or older who present for colonoscopy at White River Junction VAMC and Indiana University

Exclusion Criteria:

* includes co-morbid status of ASA III or higher, Inflammatory Bowel Disease (IBD), surgical resection of the large bowel, as well as the use of anticoagulants. Finally, potential subjects who do not report a clear effluent in the most recent bowel movement will be excluded from the study.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2018-08-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of Connecticut Health Center, Farmington, Connecticut
  - Indiana University Hospital, Indianapolis, Indiana

REFERENCES:
- [Derived] Anderson JC, Kahi CJ, Sullivan A, MacPhail M, Garcia J, Rex DK. Comparing adenoma and polyp miss rates for total underwater colonoscopy versus standard CO2: a randomized controlled trial using a tandem colonoscopy approach. Gastrointest Endosc. 2019 Mar;89(3):591-598. doi: 10.1016/j.gie.2018.09.046. Epub 2018 Oct 24. PMID 30367879

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Water Infusion First | CO2 Insufflation First
Started | 60 | 61
Completed | 60 | 61
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Water Infusion First | CO2 Insufflation First | Total
Number analyzed (Participants) | 60 | 61 | 121
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.4 (7.5) | 63.4 (8.4) | 63.4 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 12 | 28
  Male | 44 | 49 | 93
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 60 | 61 | 121
Monitored anesthesia care (MAC) [Count of Participants; unit: Participants] | 35 | 35 | 70
Colonoscopy ordered for screening purposes? [Count of Participants; unit: Participants] — Number of colonoscopies performed for screening
  Participants | 17 | 21 | 38

OUTCOME MEASURES:

1. Primary Outcome: Adenoma Miss Rate
Description: Adenoma-level miss rates will be calculated as the number of additional adenomas detected during the second examination divided by the total number of adenomas detected during both examinations
Time Frame: Through procedure, an average of 1 hr
Population: Adenoma miss rate
Measure: Number; unit: adenomas missed by first exam
Units Other Than Participants: adenomas
Arm/Group | Water Infusion First | CO2 Insufflation First
Number analyzed (Participants) | 60 | 61
Number analyzed (adenomas) | 146 | 159
adenomas missed by first exam | 52 | 37

2. Secondary Outcome: Patient-level Miss Rate
Description: Patient-level miss rates will be calculated as the number of patients with one or more adenomas detected during the second examination, divided by the total number of patients with at least one adenoma in either examination
Time Frame: 1 hour or the duration of the procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Water Infusion First | CO2 Insufflation First
Number analyzed (Participants) | 60 | 61
Participants | 27 | 23

3. Secondary Outcome: Adenoma < 6mm Detection Rate
Description: Adenoma-level miss rates will be calculated as the number of additional adenomas < 6 mm detected during the second examination divided by the total number of adenomas< 6 mm detected during both examinations.
Time Frame: 1 hour or the duration of the procedure
Population: Adenomas < 6 mm
Measure: Count of Units; unit: Adenomas < 6 mm
Units Other Than Participants: Adenomas < 6 mm
Arm/Group | Water Infusion First | CO2 Insufflation First
Number analyzed (Participants) | 60 | 61
Number analyzed (Adenomas < 6 mm) | 109 | 128
Adenomas < 6 mm | 45 | 36
Statistical Analysis 1: Comparison: Water Infusion First vs CO2 Insufflation First; Test type: Other; p = 0.48, Chi-squared

ADVERSE EVENTS:
Time Frame: As per clinical care of patient having colonoscopy, up to 30 days post procedure
Arm/Group | Water Infusion First | CO2 Insufflation First
All-Cause Mortality (participants affected / at risk) | 0/60 | 0/61
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/61
Other Adverse Events (participants affected / at risk) | 0/60 | 0/61

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-23): https://cdn.clinicaltrials.gov/large-docs/17/NCT03231917/Prot_SAP_000.pdf